

كلية طب الأسنان لجنة أخلاقيات البحث العلمي (FDASU-REC)

# الموافقة المستنيرة

| اسم المريض: | السن: | النوع: |
|-------------------|------------|--------|
| العنوان: | | |
| التليفون: محمول: | | |
| اسم ولى الأمر:درج | ة القرابة: | |

- عنوان البحث: مقارنة تاثير الادوية الطبيعية والصناعية المختلفة المستخدمه كادوية داخل قناه اللب على علاج التهاب تحت جذر السن في حالات فشل علاج اللب (تجربة إكلينيكية بالانتقاء العشوائي)
- الخلفية العلمية: يوجد عوامل عديدة يرجع لها فشل علاج اللب اهمها المسببات الميكروبية التي تتقسم الي ميكروبات هوائية ولاهوائية مثل التي تتحمل اقسي الظروف المحيطة بها وتتلائم مع اقل مصادر للغذاء والنمو . ولذالك مع التحضيرالقناه باستخدام الأدوات اللبية وتعقيمها بالمواد المضادة للميكروبات تظل انواع من البكتريا المقاومه في الاماكن الضيقة في القناه اللبية مثل القنوات الفرعية . لهذا السبب يستخدم ادوية موضعية داخل القناه اللبية بين الجلسات ولكن الانواع التقليدية مثل هيدروكسيد الكالسيوم لاتؤثر جيدا علي البكتريا المقاومة . ولذالك استخدام انواع اخري يكون لها تأثير جيد علي انواع البكتريا المختلفة الموجودة في القناه اللبية التي فشل علاجها بالادوية التقليدية هذة الانواع مثل خليط المضاد المختلفة الموجودة الالتهاب وقد استخدمت من قبل ولكن كل دواء بمفرده ووجد لها تأثير جيد . كما ان الاتجاه الجديد نحو الادويه الطبيعية مثل الكركم وقد وجد لها تأثير ممتاز علي البكتريا المقاومه الموجودة في القنوات اللبية التي فشل علاجها من قبل. ولكن وجد ان الكركم العادي له بعض العيوب مثل قلة الذوبان والانتشار وسرعة التحلل والتكسير لذالك الاتجاه نحواستخدام الكركم النانو اصبح له اهمية كبيره لانه والانتشار وسرعة العوب.
- الهدف من إجراء البحث: مقارنة كفاءه الكركم العادي والكركم النانو بخليط المضاد الحيوي ومضاد الالتهابات كادوية موضعية داخل القناه اللبية في حالات فشل علاج اللب وتقييم تاثير هم كمضادات للبكتريا وعلى تقليل الالم وايضاعلى شفاء الاتهاب تحت جذر السن.
  - مكان البحث: عيادة علاج الجذور كلية طب اسنان -جامعه عين شمس مصر
  - عدد المشاركين في البحث: ٨٠ يتم تقسيمهم الى اربعه مجموعات كل مجموعه ٢٠
    - أسلوب اختيار المشاركين في البحث:
- معايير الضم: المرضي المشاركون في البحث يجب ان لا يعانون من اي امراض صحية واعمارهم تتراوح بين ٢٠ ٦٠ سنة وقادرين علي الفهم والاستيعاب والامضاء علي الموافقة المستنيره ولديهم سنه امامية او ضاحكه بجذر واحد تم عمل لها علاج للب وفشل وتحتاج الي اعادة علاج اللب حيث يوجد التهاب تحت جذر السن
  - معايير الاستبعاد: المرضي الذين يعانون من امراض مزمنه لديهم اسنان شديدة الكسر وغير صالحه لعزلها من اللعاب وبالتي غير صالحة لاعادة علاج اللب الاسنان التي يوجد لديها علي سبيل المثال مبرد علاج اللب مكسور او ثقب تم حدوثه في علاج اللب السابق المرضى الذين لديهم تاريخ بحصولهم على اي مضادات حيوية خلال شهر قبل بدا الدراسة



#### كلية طب الأسنان

#### لجنة أخلاقيات البحث العلمى (FDASU-REC)

الاسنان التي يوجد لديها التهابات لثوية شديدة وجيوب لثوية عمقها اكثر من ٤ مم

• تفاصيل خطوات البحث: سوف يتم تقسيم ٨٠ سنه ذات قناة واحدة الي اربع مجموعات: مجموعه ١: بعد تنظيف القناه اللبية وتنشيفها يتم وضع الكركم النانو لمدة اسبوع مجموعه ٢: بعد تنظيف القناه اللبية وتنشيفها يتم وضع الكركم العادي لمدة اسبوع مجموعه ٣: بعد تنظيف القناه اللبية وتنشيفها يتم وضع خليط المضاد الحيوي (سيبر وفلوكساسين) مع مضاد الالتهابات (بروفين) لمدة اسبوع

مجموعه ٤ (مجموعة ضابطه): بعد تنظيف القناه اللبية وتنشيفها يتم وضع هيدروكسيد الكالسيوم (ميتابيست)لمدة اسبوع

يتم وضع هذة الادوية الموضعية بعد از اله حشو اللب القديم بين الجلسات ثم از التها بعد اسبوع من وضعها وبعد ذالك يتم حشو اللب من جديد ويتم تقييم تاثير كل دواء موضعي من الناحية الميكروبيولوجية وتاثيره علي تقليل الالم بين الجلسات ومتابعه الاسنان لمدة ٦ اشهر سريريا واشعاعيا لمقارنه ايضا تاثير كل دواء موضعي على شفاء الاتهاب تحت جذر السن

- عدد الزيارات المطلوبة من المتطوع و مواعيدها: ٥ زيارات كالاتي الزيارة الاولي بداية الشغل
  الزيارة الثانية بعد اسبوع من الاولي ، الزيارة الثالثه بعد شهر ، الزيارة الرابعه بعد ٣ اشهر والزيارة الاخيرة بعد ٦ اشهر.
  - اجمالي الفترة الزمنية المطلوبة من المتطوع: ٦ اشهر

المخاطر/ الأعراض الجانبية المحتمل حدوثها من إجراء البحث: لايوجد اعراض جانبية للادوية الموضعية موضوع الدراسة ولكن هناك احتمال حدوث مضاعفات مثل انفصال جزء من مبرد علاج اللب، حدوث ثقب في قناه علاج اللب، انسداد لقناه اللب، عدم التئام الكامل للالتهاب تحت جذر السن، احتمال حدوث عدوي بكتيرية بعد العلاج وعند حدوثها يتم إعطاء المريض مضاد حيوي او قد يحدث الم بعد العلاج، ومن المحتمل أيضا حدوث تورم مؤقت بعد إعادة علاج اللب، احتمال أيضا حدوث تفاعل من غسول قناه اللب (هيبوكلوريد الصوديوم) اذا تم استخدامه بضغط، عند حشو اللب قد يحدث امتداد اكثر من المعتاد للحشو علاج اللب او المادة اللاصقة للحشو تحت جذر السن.

# • الفوائد المتوقعة من البحث:

- النفقات التي سوف يتحملها المريض: لايتحمل المريض اي تكاليف
  - النفقات التي سوف يتحملها الباحث: يتحمل الباحث جميع التكاليف
- الفوائد المباشرة للمشارك المتطوع: يقلل له الالم ويزيل الالتهاب تحت جذر السن ويحصل علي العلاج الكامل للسن مجانا بدون تحمل اية تكاليف
- الفوائد العامة الغير مباشرة من البحث (الإفادة العلمية): عند نجاح احد الادوية الموضعية موضع الدراسة في تقليل الالم وتقليل البكتيريا وازاله الالتهاب تحت جذر السن يتم استخدامه على المجتمع ويصبح مادة متاحه للجميع باستخدمها لان الشركات سوف تتنافس على انتاجها وبتالي سوف يقل سعرها وبذالك ايضا سوف يتم اضافه مادة جديدة مثل الكركم النانو الي قائمة المواد الموضعية المستخدمه في علاج اللب او اعادة علاج اللب.
- التعويضات في حالة حدوث مخاطر: في حالة حدوث اي مخاطر يتم تعويض المريض بعلاجه علي نفقه الباحث ايضا حتى يتم شفاءه تماما
- البدائل المتاحة: في حالة رفضك الإشتراك في هذا البحث ستتلقى علاجك المعتاد بدون عقوبة أو خسارة أي مزايا



### كلية طب الأسنان

### لجنة أخلاقيات البحث العلمي (FDASU-REC)

• سرية معلوماتك: سوف تعامل معلوماتك بسرية كاملة و لن يطلع على بياناتك سوى الباحث الرئيسى. بعد إنتهاء الدراسة سيتم إبلاغك بنتائج البحث كما سيتم إبلاغك بأى نتائج تتعلق بحالتك الصحية.

• حقك في الإنسحاب: من حقك الإنسحاب من البحث في اي وقت دون إبداء أسباب دون أي عواقب سلبية عليك.

• عند وجود أى إستفسار لديك يمكنك الإتصال ب:

اسم الباحث الرئيسي: طبيب/ روضه محمد عبد الرحمن بغدادي التليفون: ١١٤٢٣٦١٠٧٤.

اسم المشرف الرئيسي: ١.د. كريم مصطفى البطوطي

من ينوب عنه: د/ سارة حسام فهمي التايفون:

مقرر لجنة الأخلاقيات: أ.م.د/ مارى مدحت التليفون: 01222892635



كلية طب الأسنان لجنة أخلاقيات البحث العلمي (FDASU-REC)

| لعت و فهمت الإجراءات التي ستتم من خلال هذا البحث و وافقت عليها | ر اىنى اطك | ۱عر |
|---|---|---|
|---|---|---|

المشارك في البحث:

الأسم:

التوقيع (البصمة):

الشاهد الأول (ان وجد/ في حالة الموافقة الشفهية):

الشاهد الثاني (ان وجد/ في حالة الموافقة الشفهية):

التاريخ:

إقرار الطبيب المشرف/ الباحث الرئيسى على البحث: روضة محمد عبد الرحمن بغدادي أتعهد بالحفاظ على سرية المعلومات الخاصة يالشخص محل البحث توقيع الطبيب المشرف:

التاريخ:

## ملحوظة<u>:</u>

- 1. من حق المتطوع الانسحاب من البحث في أي وقت
  - 2. يجب حصول المتطوع على صورة من الإقرار
- قب إجازة خطوات هذاً البحث من الناحية العلمية والأخلاقية من قبل المختصين بكلية طب الأسنان جامعة عين شمس
  في / / بعد التأكد من أن البحث يتوافق مع الميثاق الاخلاقي للكلية ، وان الفائدة المرجوة منه تربو على المخاطر المحتملة
  - 4. رقم مسلسل الموافقة